CLINICAL TRIAL: NCT05192980
Title: SIOPEN BIOPORTAL, An International Registry Linked to a Virtual Biobank for Patients With Peripheral Neuroblastic Tumours
Acronym: BIOPORTAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2020-17
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma; Ganglioneuroblastoma; Ganglioneuroma
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroblastoma; Ganglioneuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral neuroblastic tumors (ganglioneuroma, ganglioneuroblastoma and neuroblastoma) (Other)
  Interventions: Other: No Intervention NA

INTERVENTIONS:
Other: No Intervention NA — Additional blood sampling (not mandatory)
  Other Names: Bio-sampling

SUMMARY:
The SIOPEN BIOPORTAL is a prospective non-therapeutic multi-centre international study aimed at developing an international Registry linked to a Virtual Biobank for all the patients with peripheral neuroblastic tumor within countries of the SIOPEN network. The overall aim of this study is to provide a GDPR-compliant framework to collect basic clinical annotations, biological and genetic features and information about the location on biospecimens for all the patients with a peripheral neuroblastic tumor including neuroblastoma, ganglioneuroblastoma and ganglioneuroma in the SIOPEN network.

This study will support data and sample management and intensify cross-borders data and sample sharing fostering translational and clinical research. The post-hoc hypothesis formulated based on the data generated in this study will be used as statistical basis for future precision medicine programs based on improved biological characterization, patient stratification and therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

I-1. Patients with PNT: ganglioneuroma or ganglioneuroblastoma or neuroblastoma, I-2. At the time of initial diagnosis of neuroblastic tumour, or at relapse/progression if not yet registered I-3. Written patient informed consent, or parents or legal representative written informed consent and assent of the child, adolescent or young adult

Non-Inclusion Criteria:

R-1. (Adult) Patients with olfactory neuroblastoma R-2. Central nervous system (CNS) neuroblastoma (as per the WHO classification)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2038-11-02 (Estimated); Study Completion 2038-11-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients having their clinical data registered | 6 months
  Registry Outcome: Rate of patients having their clinical data registered throughout their treatment and follow-up from the total of patients registered
Rate of patients for whom information on biological samples/material is collected | 6 months
  Virtual Biobank Outcome: Rate of patients for whom information on biological samples/material collected and stored in SIOPEN is available from the total of patients registered

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  Investigation of the impact of the variables currently used for assignment to risk groups and treatment stratification (MYCN Status, ALK Status, stage, age, primary tumor site) on progression-free survival (PFS) using the Kaplan-Meier method
Overall-survival (OS) | 12 months
  Investigation of the impact of the variables currently used for assignment to risk groups and treatment stratification (MYCN Status, ALK Status, stage, age, primary tumor site) on overall-survival (OS) using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Locations (38):
- Fakultni nemocnice v Motole, Prague, Czechia
- France (27):
  - CHU Amiens, Amiens
  - Chu Angers, Angers
  - Hôpital Jean Minjoz, Besançon
  - Hôpital des enfants, Bordeaux
  - Chru Brest, Brest
  - CHU CAEN - Fédération de cancérologie - niveau 21, Caen
  - CHU D'Estaing de CLERMONT FERRAND, Clermont-Ferrand
  - DIJON Hôpital d'enfants, Dijon
  - Chu Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital d'Enfants de la Timone, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Chr Nantes, Nantes
  - CHU NICE, Nice
  - Institut Curie, Paris
  - Hôpital Armand Trousseau, Paris
  - Hôpital Jean Bernard, Poitiers
  - Chu Reims, Reims
  - Chu Hopital Sud, Rennes
  - Hôpital Charles NICOLLE, Rouen
  - Hôpital Nord, Saint-Etienne
  - Hôpital Hautepierre-CHU Strasbourg, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Hôpital Clocheville, Tours
  - CHU NANCY- Hôpital d'Enfants, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Oslo Universitetssykehus, Oslo, Norway
- Switzerland (9):
  - Kantonsspital Aarau AG, Aarau
  - Universitäts-Kinderspital beider Basel UKBB, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - HUG Hôpitaux Universitaires Genève, Geneva
  - CHUV, Centre hospitalier universitaire vaudois, Lausanne
  - Kinderspital Zentralschweiz, Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Universitäts-Kinderspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://www.siopen.net/